CLINICAL TRIAL: NCT05153733
Title: Improved Implant for Reconstruction Purposes After Mandibular Resection
Acronym: RifRam
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: End point is reached with 1 implant which is removed within the observation period
Sponsor: The Netherlands Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N19IRM; NL74131.031.20 (Registry Identifier: CCMO ABR)
Record Dates: First submitted 2021-11-29; First posted 2021-12-10 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Head and Neck Cancer; Oral Cancer
Keywords: surgery; COMMANDO
MeSH Terms: conditions — Head and Neck Neoplasms; Mouth Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RIFRAM implant (Experimental): RIFRAM implant
  Interventions: Device: RIFRAM implant

INTERVENTIONS:
Device: RIFRAM implant — Participants will receive the newly developed, patient-specific RIfRaM mandibular implant.
  Other Names: COMMANDO

SUMMARY:
Study design: A single center non-randomized, prospective clinical feasibility study.

Study population: Study population is composed of 10 patients ineligible for a free-flap bone reconstruction.

Intervention: The selected patients will receive the newly developed, patient-specific RIfRaM mandibular implant.

Objective: The aim is to provide enough evidence through model analysis, physical tests and clinical study of 10 patients that our new type of personalized mandibular implant is safe to use, resulting in significantly fewer complications and can be practically placed during the surgery, without any complications.

Main study parameters/endpoints: The study endpoint is to use the RifRaM without any implant related complications and a perfect mandibular fit.

DETAILED DESCRIPTION:
The preoperative bony resection planning and the design of the RifRam implant will be carried out on 3D reconstructed CT image of the mandible. The necessary resection planes will be marked on the 3D model. This segment will be removed virtually and replaced by the designed RifRam implant. The form of the implant will follow the contours of the native healthy mandible. In case, extensive bone destruction of the mandible does not allow copying the contours, contralateral side of the mandible will be virtually mirrored and used to design the implant. The design of the implant will be carried out within the NKI/AVL and the data will be preserved in restricted access folders. The designed implant will be printed with a hollow mesh core by Mobius. A matching cutting guide will be printed as well. Two copies of the implant will be delivered in case one would be accidentally be unsterile (see 5.3). The cutting guides are used to cut the mandible at exactly the intended places. The implant and the cutting guide will be delivered to the hospital and sterilized by Clinium for clinical use.

The patient will undergo a COMMANDO (combined mandibulectomy and neck dissection) procedure. The steps of this procedure are well defined and can be found in iProva. The oncological resection will be carried out in the standard fashion. Mandible saw cutting guides are used as standard procedure. The patient specific mandible cutting guide will be fixed on the mandible and the cuts to the mandible will be made through the cutting slots. This step enables that the mandible defect matches exactly the RifRam implant. After the resection is completed and the surgical site irrigated as per standard procedure, the Rifram implant will be placed to fill the bone defect. The implant will be fixed with 2.7 mm locking screws produced by KLS Martin. These screws are used are used as standard and are available in stock in the operation complex. The soft tissue defect will be reconstructed using a regional flap such as pectoralis major musculocutaneous flap. The rest of the procedure will be completed as per established clinical protocol.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years at time of study entry.
* T4 oral cavity tumor with mandible invasion, requiring segmental mandibulectomy.
* Reconstruction with free fibula flap not feasible because of any or a combination of the following reasons:

oCT angiography of the legs and/or the neck shows severe stenosis of the ves-sels.

* Previous medical history of severe atherosclerotic disease.
* General health condition necessitating a shorter operation time.

  * Cases will be discussed in the multidisciplinary tumor board that they are eligible for composite resection but not eligible for free fibula flap.
  * Written informed consent.

Exclusion Criteria:

* Patients who are eligible for free fibula flap.
* Pregnancy.
* General health condition does not allow surgery
* History of psychiatric disability judged by the investigator to potentially hamper compliance with the study protocol and follow-up schedule.
* Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2021-11-29 (Actual); Primary Completion 2024-03-13 (Actual); Study Completion 2024-03-13 (Actual)

PRIMARY OUTCOMES:
Surgical fit | intra-operative
  good fit during surgery, suboptimal fit of the mandible making placement not possible.
Complications | implant loss in 1-year post-operational follow-up.
  Implant related complications leading to implant loss

CONTACTS AND LOCATIONS:
Overall Officials: Baris Karakullukcu, PhD, Principal Investigator — The Netherlands Cancer Institute
Locations (1):
- Antoni van Leeuwenhoek, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No